CLINICAL TRIAL: NCT02719795
Title: Pectoral Nerves Blocks and Their Effect on Chronic Pain After Breast Cancer Surgery
Brief Title: Pectoral Nerves Blocks for Chronic Pain
Acronym: PNBCP
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XJTU1AF-CRS-2016-003
Record Dates: First submitted 2016-03-15; First posted 2016-03-25 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2016-04

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasms; Nerve block; Anesthesia
MeSH Terms: conditions — Breast Neoplasms | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine (Experimental): Ropivacaine hydrochloride injection； Generic name：Naropin； Dosage form：Liquid、Injectable formulation； Dosage：105mg；30ml； Frequency：Once.
  Interventions: Drug: Ropivacaine
- Normal saline (Placebo Comparator): Medical Normal saline Generic name：Normal saline； Dosage form：Liquid、Injectable formulation； Dosage：30ml； Frequency：Once.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ropivacaine — Local injection of local anesthetic into the fascial spaces
  Other Names: Naropin
  Arms: Ropivacaine
Drug: Normal saline — Sodium chloride solution commonly used in clinical which equal to human plasma osmotic pressure.
  Other Names: Stroke-physiological saline solution
  Arms: Normal saline

SUMMARY:
The purpose of this study is to determine whether pectoral nerves blocks（PECS） would reduce chronic pain at 3 months after modified radical mastectomy（MRM）surgery.

DETAILED DESCRIPTION:
One hundred and forty adult female participants scheduled for elective unilateral modified radical mastectomy under general anesthesia are randomly allocated to receive either general anesthesia plus Pecs block(Pecs group, n=70) or general anesthesia alone (control group, n=70).

After arrived in the operating room，the participants in the control group are accepted the general anesthesia.Whereas，after anesthesia induction，the participants in the Pecs group receive an ultrasound-guided Pecs block and a 15 minute observation time prior before the start of the operation.

Pecs block technology： A broadband (5-12 hertz) linear array probe of Sonosite Edge portable ultrasound system (Sonosite Inc,Bethel,Washington) is used, with an imaging depth of 4 to 6 cm. After cleaning the infraclavicular and axillary regions with chlorhexidine, the probe is placed below the lateral third of the clavicle, similar to what is done when performing infraclavicular brachial plexus block. After recognition of the appropriate anatomical structures, the skin puncture point is infiltrated with 2% lignocaine, then the block is performed by using a 20-gauge Tuohy needle. The needle is advanced to the tissue plane between the pectoralis major and pectoralis minor muscle at the vicinity of the pectoral branch of the acromiothoracic artery, and 10 mL of 0.35% ropivacaine deposited. In a similar manner, 20 mL is deposited at the level of the third rib below the serratus anterior muscle with the intent of spreading injectate to the axilla.

ELIGIBILITY:
Inclusion Criteria:

* Modified radical mastectomy
* American Society of Anesthesiologists physical status 1-3
* BMI 18-35 kg/m2

Exclusion Criteria:

* Declining to give written informed consent；
* Uncontrolled hypertension；
* Allergy to local anesthetics；
* Pregnancy；
* Alcohol or drug abuse；
* Prior breast surgery except for diagnostic biopsies；
* Contraindication to the use of regional anesthesia；
* History of chronic pain or psychiatric disorder and pregnant patients；
* Consumption of NSAID, cyclooxygenase-2 inhibitors or paracetamol within 24 hours before the investigation；
* Infection at the needle site.
* Inability to properly describe postoperative pain to investigators (eg, language barrier, neuropsychiatric disorder)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
The incidence of chronic postoperative pain for 3 months after modified radical mastectomy surgery | 3 months after modified radical mastectomy surgery
  An anesthesiologist interviews the patients by phone to determine the postoperative pain at 3 months after surgery. Chronic pain is defined as pain in the surgical area or the ipsilateral arm, present at least 4 days a week, with an intensity of 3 or more on the verbal rating scale（0=no pain to 10=worst imaginable pain),described as a typical neuropathic pain consisting of burning pain, shooting pain, pain evoked by pressure, and deep blunt pain.

SECONDARY OUTCOMES:
Postoperative Numerical Rating scale (NRS) score for pain | 0 hour postoperative
  Pain scores（0-10）during rest and cough based on measurement at 0 hour postoperative.
Postoperative Numerical Rating scale (NRS) score for pain | 4 hours postoperative
  Pain scores（0-10）during rest and cough based on measurement at 4 hours postoperative.
Postoperative Numerical Rating scale (NRS) score for pain | 12 hours postoperative
  Pain scores（0-10）during rest and cough based on measurement at 12 hours postoperative.
Postoperative Numerical Rating scale (NRS) score for pain | 24 hours postoperative
  Pain scores（0-10）during rest and cough based on measurement at 24 hours postoperative.
Postoperative Numerical Rating scale (NRS) score for pain | 48 hours postoperative
  Pain scores（0-10）during rest and cough based on measurement at 48 hours postoperative.
Postoperative Numerical Rating scale (NRS) score for pain | 72 hours postoperative
  Pain scores（0-10）during rest and cough based on measurement at 72 hours postoperative.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hosipital of Xi'an Jiaotong Univercity, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Amaya F, Hosokawa T, Okamoto A, Matsuda M, Yamaguchi Y, Yamakita S, Taguchi T, Sawa T. Can acute pain treatment reduce postsurgical comorbidity after breast cancer surgery? A literature review. Biomed Res Int. 2015;2015:641508. doi: 10.1155/2015/641508. Epub 2015 Oct 1. PMID 26495309
- [Result] Oeffinger KC, Fontham ET, Etzioni R, Herzig A, Michaelson JS, Shih YC, Walter LC, Church TR, Flowers CR, LaMonte SJ, Wolf AM, DeSantis C, Lortet-Tieulent J, Andrews K, Manassaram-Baptiste D, Saslow D, Smith RA, Brawley OW, Wender R; American Cancer Society. Breast Cancer Screening for Women at Average Risk: 2015 Guideline Update From the American Cancer Society. JAMA. 2015 Oct 20;314(15):1599-614. doi: 10.1001/jama.2015.12783. PMID 26501536
- [Result] Bolin ED, Harvey NR, Wilson SH. Regional anesthesia for breast surgery: Techniques and benefits. Current Anesthesiology Reports 2015;5:217-224.
- [Result] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Result] Poleshuck EL, Katz J, Andrus CH, Hogan LA, Jung BF, Kulick DI, Dworkin RH. Risk factors for chronic pain following breast cancer surgery: a prospective study. J Pain. 2006 Sep;7(9):626-34. doi: 10.1016/j.jpain.2006.02.007. PMID 16942948
- [Result] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Result] Jung BF, Ahrendt GM, Oaklander AL, Dworkin RH. Neuropathic pain following breast cancer surgery: proposed classification and research update. Pain. 2003 Jul;104(1-2):1-13. doi: 10.1016/s0304-3959(03)00241-0. No abstract available. PMID 12855309
- [Result] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Result] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Result] Perez MF, Miguel JG, de la Torre PA. A new approach to pectoralis block. Anaesthesia. 2013 Apr;68(4):430. doi: 10.1111/anae.12186. No abstract available. PMID 23488849
- [Result] Perez MF, Duany O, de la Torre PA. Redefining PECS Blocks for Postmastectomy Analgesia. Reg Anesth Pain Med. 2015 Nov-Dec;40(6):729-30. doi: 10.1097/AAP.0000000000000243. No abstract available. PMID 26488081
- [Result] Ibarra MM, S-Carralero GC, Vicente GU, Cuartero del Pozo A, Lopez Rincon R, Fajardo del Castillo MJ. [Chronic postoperative pain after general anesthesia with or without a single-dose preincisional paravertebral nerve block in radical breast cancer surgery]. Rev Esp Anestesiol Reanim. 2011 May;58(5):290-4. doi: 10.1016/s0034-9356(11)70064-0. Spanish. PMID 21692253
- [Result] Karmakar MK, Samy W, Li JW, Lee A, Chan WC, Chen PP, Ho AM. Thoracic paravertebral block and its effects on chronic pain and health-related quality of life after modified radical mastectomy. Reg Anesth Pain Med. 2014 Jul-Aug;39(4):289-98. doi: 10.1097/AAP.0000000000000113. PMID 24956453
- [Result] Vilholm OJ, Cold S, Rasmussen L, Sindrup SH. The postmastectomy pain syndrome: an epidemiological study on the prevalence of chronic pain after surgery for breast cancer. Br J Cancer. 2008 Aug 19;99(4):604-10. doi: 10.1038/sj.bjc.6604534. PMID 18682712